CLINICAL TRIAL: NCT01010958
Title: A Pilot Study of Adjuvant Valproate for Patients With High Grade Sarcomas
Brief Title: Adjuvant Valproate for High Grade Sarcomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Kevin Kalinsky, Assistant Professor of Clinical Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAD4523
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: High Grade Sarcoma
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valproate (Experimental): Valproic Acid taken orally, daily to reach serum levels between 50 to 100 µg/mL.
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid — Subjects should initiate therapy at 10 to 15 mg/kg/day. The dosage should be increased by 5 to 10 mg/kg/week to achieve optimal clinical response. Optimal clinical response is achieved at daily doses below 60 mg/kg/day. If satisfactory clinical response has not been achieved, plasma levels should be measured to determine whether or not they are in the usually accepted therapeutic range (50 - 100 µg/mL).
  Other Names: Depakene

SUMMARY:
For patients initially presenting with localized sarcoma the standard of care is surgery followed by with radiation therapy (if feasible). Subsequent or adjuvant cytotoxic based chemotherapy even for aggressive sarcoma histopathologies (as commonly done for colorectal cancer or breast cancer) is controversial since over 20 individual adjuvant randomized clinical trials have not been able to consistently demonstrate a statistically significant improvement in overall survival. Maturation or differentiation therapy provides an opportunity to fundamentally change the biology of the underlying cancer (and thus its overall prognosis) by promoting cellular maturation within that cancer. A change from a poorly 'differentiated/high grade' tumor to a well 'differentiated/low grade' tumor is attainable and can change an individual's median time of survival from months to decades. The investigators have significant preclinical data that differentiation therapy using a group of drugs referred to as histone deacetylase inhibitors (such as Valproate, also a commonly used and safe anti seizure medication) is feasible for sarcomas. This approach has not been clinically addressed in solid tumors. Since adjuvant therapy is controversial for sarcomas, and building on the investigators' preclinical data, adjuvant based differentiation therapy using valproate would be predicted to be both safe and potentially extremely beneficial in terms of a) increasing the time to disease recurrence, b) improving the histology upon recurrence; and c) improving overall survival in patients with sarcomas.

Patients with high grade sarcomas will receive Valproate in the adjuvant setting daily and clinically/radiologically followed until recurrence. Relapse free survival, time to local failure, time to distant failure, overall survival, and comparative histopathology of primary and recurrence will be assessed.

DETAILED DESCRIPTION:
Adjuvant chemotherapy for high grade soft tissue sarcomas is controversial. Given the fact that approximately 50% of patients receiving optimum treatment will recur in three years and die of recurrence within five years, smarter adjuvant options are needed. One such treatment option would be to "differentiate" the high grade sarcoma into a low grade sarcoma upon recurrence. This differentiation effect will reduce the risk of subsequent death by 50% as determined by the overall survival difference between high grade/poorly differentiated and low grade/ well differentiated sarcomas. Given that differentiation takes place on a time scale that is significantly longer than cytotoxic effects, the optimum time to initiate differentiation therapy is in the adjuvant setting; when the time to disease recurrence is measured in months to years.

The histone deacetylase inhibitor, Valproate, has been shown to promote differentiation in myeloid malignancies when administered in standard dosing regiments. We have recently shown that sarcomas are conceptually similar to hematopoietic malignancies, in that both represent diseases of aberrant development in which developing cells along their respective lineages arrest and transform at various points of differentiation. We have recently shown in vitro that, as for acute promyelocytic leukemia, sarcomas can be reprogrammed to reenter normal differentiation via epigenetic modulation using histone deacetylase inhibitors. It is therefore appealing to study Valproate based differentiation therapy in the adjuvant setting for sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed high-grade soft tissue sarcoma. Patients may be entered based on local pathology.
* Surgical paraffin tissue (preferable) and/or 10-15 unstained slides must be available for baseline analysis.
* No evidence of measurable disease.
* Primary surgery no longer than 12 weeks prior to starting treatment or within 4 weeks of completing adjuvant cytotoxic chemotherapy, if administered.
* No more than four cycles of adjuvant based chemotherapy.
* No active liver disease.
* Are 18 years of age or older.
* Have a life expectancy greater than 3 months.
* Have an ECOG performance status of 0 or 1.
* Is capable of providing voluntary written informed consent in accordance with all applicable regulations and follow the study procedures. Patients must be capable of understanding the investigational nature, potential risks and benefits of the study.

Exclusion Criteria:

* Have inadequate organ function at the screening visit as defined by the following laboratory values: platelet count less than 100 x 109/L; hemoglobin less than 9.0 g/dL; absolute neutrophil count (ANC) less than 1.5 x 109/L; international normalized ratio (INR) greater or equal to 1.5 and a PTT greater than the upper limit of normal (ULN) within 1 week prior to randomization; creatinine clearance (Cockroft Gault) less than 50ml/min; urine protein: creatinine ratio greater or equal to 1.0 at screening; aspartate transaminase (AST) greater than 1.5 x ULN; alanine transaminase (ALT) greater than or equal to 1.5 x ULN; total bilirubin greater than 1.5 x ULN or greater or equal to 5 x ULN in patients with liver metastases.
* Prior history of valproate use.
* History or active liver disease.
* Evidence of bleeding diathesis or coagulopathy.
* Has uncontrolled active systemic infection requiring therapy.
* Have had treatment for a cancer other than sarcoma within 5 years prior to enrollment, with the exception of basal cell carcinoma or cervical cancer in-situ.
* Have known human immunodeficiency virus (HIV) positive or hepatitis B surface antigen positive status or known active hepatitis C infection. Patients assessed by the investigator to be at risk for HIV, hepatitis B or C infection should be tested in accordance with local regulations.
* Are a pregnant or breast feeding female. Confirmation that the patient is not pregnant must be established by a negative serum beta human chorionic gonadotropin (beta hCG) pregnancy test result obtained during the Screening Period. Pregnancy testing is not required for postmenopausal or surgically sterilized women.
* Are unwilling to employ adequate means of contraception (condoms, diaphragm, birth control pills, injections, intrauterine device, or abstinence).
* Has a serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Female subjects must either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of lower grade sarcoma | Up to 3 years
  The primary end point will be evaluated by the 3-year recurrence rate of lower grade sarcoma histopathologically (or more well differentiated as compared to the primary tumor) amongst those who experience 3-year sarcoma recurrence.

SECONDARY OUTCOMES:
Relapse free survival rate | Up to 3 years
Time to local failure | Up to 3 years
Time to distant failure | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kalinsky, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States